CLINICAL TRIAL: NCT06839209
Title: Pilot Study to Evaluate Advantages and Disadvantages of TOXCLEAN As Add on Treatment to SOC in Patients with Clostridium Difficile-associated Diarrhea
Brief Title: Advantages and Disadvantages of TOXCLEAN As Add on Treatment to SOC in Patients with Clostridium Difficile-associated Diarrhea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ABResearch S.r.l. (Industry)
Collaborators: Nextrasearch S.r.l.s. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TOXCCAD
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Clostridium; Difficile, As Cause of Disease Classified Elsewhere; Clostridium Difficile Diarrhea
Keywords: clostridium difficile; clostridium; cdad

STUDY DESIGN:
Intervention Model Description: Cohort A: 1 g of Toxclean once a day for 28 days plus SoC therapy Cohort B: 1 g of Toxclean twice daily for 28 days plus SoC therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single dosage (Experimental): 1 g of Toxclean once a day for 28 days plus SoC therapy
  Interventions: Device: Toxclean 1g
- Double dosage (Experimental): 1 g of Toxclean twice daily for 28 days plus SoC therapy
  Interventions: Device: Toxclean 1g

INTERVENTIONS:
Device: Toxclean 1g — 1 g of Toxclean once or twice daily for 28 days

SUMMARY:
This is a single center, randomized, exploratory clinical investigation that will evaluate the safety and efficacy of Toxclean (ABResearch srl) as add on treatment to Standard therapy in 24 patients with recurrent CDAD.

Eligible subjects will be adult patients with recurrent CDAD. Recurrent CDAD, for the purpose of this protocol, is defined as one or more new episode of diarrhea (Ned) within two months from the end of the SoC treatment. The objective of this pilot study is to evaluate whether 1 or 2 grams of Toxclean powder is orally administrable and well tolerated as add on treatment to SoC in patients with recurrent CDAD.

DETAILED DESCRIPTION:
This is a single center, randomized, exploratory clinical investigation that will evaluate the safety and efficacy of Toxclean (ABResearch srl) as add on treatment to Standard therapy in 24 patients with recurrent CDAD.

Eligible subjects will be adult patients with recurrent CDAD. Recurrent CDAD, for the purpose of this protocol, is defined as one or more new episode of diarrhea (Ned) within two months from the end of the SoC treatment. The objective of this pilot study is to evaluate whether 1 or 2 grams of Toxclean powder is orally administrable and well tolerated as add on treatment to SoC in patients with recurrent CDAD. Primary

* Percentage of patients that complete Toxclean schedule treatment; Secondary
* Safety and tolerability of two different dosage of oral Toxclean treatment;
* Reduction of toxin amount in fecal sample;
* Clinical response after 28-day oral administration of two different dosage of TOXCLEAN in combination with SoC therapy;
* CDAD symptoms improvements during treatment and follow up periods;
* Fecal concentration of Toxclean;

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, male or female, at the time of informed consent
* Signed informed consent by patient, or where applicable, patient's legally authorized representative;
* Diagnosis of recurrent CDAD, defined as those episodes of C. Difficile associated diarrhea occurring 2-8 weeks after either the symptoms resolution of a previous CDAD episode or C. difficile negativization of fecal sample.
* Detection of C. difficile toxins by nucleic acid amplification tests (NAAT), EIA or GDH;
* Received at least one course of adequate antibiotic therapy for CDAD (≥ 10 days of vancomycin at a dose of ≥125 mg four times per day, ≥ 10 days of metronidazole at a dose of 500mg three times per day or fidaxomixin 200mg twice a day for 10 days)

Exclusion Criteria:

* History of C. difficile complicating inflammatory bowel disease (Crohn's disease, ulcerative colitis), or history of bowel resection surgery (other than uncomplicated appendectomy) or history of other infectious diarrhea or diarrhea of unknown etiology since the initial episode of CDAD;
* Participants who require oral anticoagulant medications, including but not limited to warfarin and NOACs (novel oral anticoagulants);
* Major gastrointestinal surgery within 3 months of enrollment;
* History of swallowing difficulties, including dysphagia or odynophagia for liquids or solids;
* Clinically immunocompromised due to any primary immune or autoimmune deficiency, as a result of chronic disease, cancer or medication used to treat these diseases
* Consumption of the following prescription medications during the current enrollment episode: Bezlotuxamab/Zinplava Is pregnant or lactating Known hypersensitivity to the active principle or excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients that complete Toxclean schedule treatment | 28 days
  The primary objective of this early feasibility clinical study is to evaluate whether 1 or 2 grams of Toxclean powder is orally administrable and well tolerated as add on treatment to SoC in patients recurrent

SECONDARY OUTCOMES:
the assessment of the safety and tolerability of two different dosage of oral Toxclean treatment | 28 days
  Safety and tolerability of two dosage of oral Toxclean powder plus SoC assessed by number of participants who experienced adverse events
the clinical response after 14-day oral administration of two different dosage of TOXCLEAN in combination with SoC therapy; | 14 days
  time to resolution of diarrhea: time in days from start of treatment to the first formed bowel movement
the CDAD symptoms improvements during treatment and follow up periods | 2 months
  reduction of CDAD symptoms such as abdominal pain, nausea etc
Measurement of Toxclean fecal concentration of Toxclean | 28 days
  C. difficile toxins in fecal sample;

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Cammarota, Professor, Principal Investigator — Direttore U.O.C. GASTROENTEROLOGIA Policlinico Gemelli
Locations (1):
- Policlinico Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
Study report published
Supporting Information: CSR
Time Frame: After Study conclusion, no time limits
Access Criteria: Published on Peer journals